CLINICAL TRIAL: NCT02628405
Title: Phase I/II, Open-Label Study of R-ICE (Rituximab-Ifosfamide-Carboplatin-Etoposide) With Lenalidomide (R2-ICE) in Patients With First-Relapse/Primary Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: R-ICE and Lenalidomide in Treating Patients With First-Relapse/Primary Refractory Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU051417I; NCI-2015-01990 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU051417I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Carboplatin; Etoposide; Ifosfamide; Lenalidomide; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (R2-ICE) (Experimental): Patients receive lenalidomide PO daily on days 1-14, rituximab IV on day 1, ifosfamide IV over 24 hours on day 2, carboplatin IV over 1-2 hours on day 2, and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving CMR, PMR, or NMR may receive 2 more cycles per physician discretion. After completion of 2 cycles of R2ICE treatment, patients achieving objective status of CMR, PMR or NMR may proceed to SCT during the event monitoring phase.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide when given together with rituximab-ifosfamide-carboplatin-etoposide (R-ICE) and to see how well they work in treating patients with diffuse large B-cell lymphoma that has returned after a period of improvement (relapsed) and that has not responded to previous treatment (refractory). Drugs used in chemotherapy, such as rituximab, ifosfamide, carboplatin, etoposide, and lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving lenalidomide with R-ICE may be a better treatment for patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and maximum tolerated dose (MTD) of the addition of lenalidomide to the R-ICE chemoimmunotherapy regimen (lenalidomide-rituximab-ifosfamide-carboplatin-etoposide [R2ICE]) for the treatment of primary-refractory/first-relapse B-cell lymphoma. (Phase I) II. To determine if the addition of lenalidomide (based on dose determination from phase I) to the R-ICE chemoimmunotherapy regimen (R2-ICE) would lead to clinically meaningful improvement in the overall response rates (ORR) for patients with first-relapse/refractory diffuse large B-cell lymphoma (DLBCL). (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the effect of the addition of lenalidomide to RICE on the number (percentage) of patients proceeding to stem cell transplant (SCT).

II. To evaluate the effect of the addition of lenalidomide to RICE on other surrogate outcome measures including complete metabolic response (CMR) rate and overall survival.

III. To describe the toxicities associated with the addition of lenalidomide to the R-ICE chemoimmunotherapy regimen (R2ICE).

CORRELATIVE RESEARCH OBJECTIVES:

I. To evaluate ORR based on germinal center B-cell-like (GCB) versus non-GCB subtypes.

II. To evaluate ORR based on percent standardized uptake value (SUV) reduction and percent anatomic size reduction on interim positron emission tomography (PET)/computed tomography (CT) scans.

III. To evaluate ORR based on minimal residual disease (MRD) detection (positive versus [vs.] negative) and quantification after 2 cycles of treatment.

IV. Future tissue and blood based studies.

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

Patients receive lenalidomide orally (PO) daily on days 1-14, rituximab intravenously (IV) on day 1, ifosfamide IV over 24 hours on day 2, carboplatin IV over 1-2 hours on day 2, and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving CMR, partial metabolic response (PMR), or no metabolic response (NMR) may receive 2 more cycles per physician discretion. After completion of 2 cycles of R2ICE treatment, patients achieving objective status of CMR, PMR or NMR may proceed to SCT during the event monitoring phase.

After completion of study treatment, patients are followed up every 3 months for 3 years and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Phase I: Histological confirmation of expressing CD20 antigen as determined by pathology at the respective institution and central pathology review at Mayo Clinic Rochester; all types of B-cell lymphomas are allowed to participate; patients with primary mediastinal large B-cell (PMLBCL) or transformed lymphoma are allowed to participate
* Phase II: Histological confirmation of DLBCL expressing CD20 antigen as determined by pathology at the respective institution and central pathology review at Mayo Clinic Rochester; patients with primary mediastinal large B-cell (PMLBCL) or transformed lymphoma are not allowed to participate
* Measurable disease (at least 1 lesion >= 1.5 cm in diameter) as detected by PET/CT
* Only 1 line of previous anti-lymphoma therapy is allowed and not currently receiving any other agent that would be considered as a treatment for the lymphoma; patients must be >= 2 weeks from prior anti-lymphoma therapy; the use of steroids and/or rituximab up to 1 week prior to registration for management of symptoms is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Absolute neutrophil count (ANC) >= 1500/mm^3, obtained =< 7 days prior to registration
* Platelet count >= 75,000/mm^3, obtained =< 7 days prior to registration
* Total bilirubin =< 2 x upper limit of normal (ULN) (unless related to lymphoma or Gilbert's disease) OR =< 5 x ULN for subjects with documented or suspected Gilbert's disease, or related to involvement of the liver by the lymphoma, obtained =< 7 days prior to registration
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN unless evidence of the direct liver and/or bone involvement by lymphoma, then =< 5 x ULN, obtained =< 7 days prior to registration
* PHASE I: Subjects must have calculated creatinine clearance >= 60 ml/min by Cockcroft-Gault formula, obtained =< 7 days prior to registration
* PHASE II: Subjects must have calculated creatinine clearance >= 30 ml/min by Cockcroft-Gault formula, obtained =< 7 days prior to registration
* For women of childbearing potential only: Negative pregnancy test =< 10-14 days prior to registration; NOTE: the patient must have an additional negative pregnancy test =< 24 hours prior to receiving the initial prescription of lenalidomide, per requirements of the REVLIMID Risk Evaluation and Mitigation Strategies (REMS) program
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study [i.e. active treatment and observation])
* Willing to provide blood samples for correlative research purposes
* Considered transplant-eligible, as determined by the opinion of the investigator at the participating institution; the participating institution does not need to be a transplant center but patients can be referred to a transplant center if needed
* Willing and able to register into and comply with the mandatory requirements of Celgene's REVLIMID REMS program
* Females of reproductive potential are willing and able to adhere to the scheduled pregnancy testing as required by Celgene's REVLIMID REMS program
* Willing and able to take aspirin (81 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin)

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

    * NOTE: patients unwilling or unable to do any of the following are also excluded:

      * Men must agree to use a latex condom during sexual contact with a female of child-bearing potential even if they have had a successful vasectomy
      * Women of child bearing potential must agree to use 2 methods of reliable contraception simultaneously
      * All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial; patients with HIV on antiretroviral therapy other than zidovudine (AZT) and/or stavudine and without prior acquired immunodeficiency syndrome (AIDS) defining conditions and adequate CD4 count (> 400) are eligible
* History of myocardial infarction =< 180 days prior to registration or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm; patients must be >= 2 weeks from prior anti-lymphoma therapy; the use of steroids and/or rituximab up to 1 week prior to registration for management of symptoms is allowed
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: non-melanotic skin cancer, carcinoma-in-situ of the cervix, or any cancer that, in the judgment of the investigator, has been treated with curative intent and will not interfere with the study treatment plan and response assessment; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment such as radiation, chemotherapy, or immunotherapy for their cancer
* Unable or unwilling to take any prophylaxis; patients with history of or new/active deep vein thrombosis/embolism/thrombophilia are allowed to participate if they are on appropriate therapeutic anticoagulation during the treatment on the trial; these patients would not need the aspirin with the lenalidomide unless clinically indicated; therefore, patients must be able and willing to receive anticoagulation (prophylaxis versus therapeutic as clinically indicated)
* History of radiation therapy to >= 25% of the bone marrow for other diseases
* Receiving erythroid stimulating agents (epoetin alfa [EPO]: Procrit, Aranesp)
* Patients with active or prior central nervous system (CNS) lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells; NOTE: these patients are usually treated with CNS directed therapy; screening for cerebrospinal fluid (CSF)/CNS involvement is NOT required but can be performed per treating medical doctor (MD) discretion
* Active hepatitis B as defined by seropositivity for hepatitis B surface antigen (HBsAg); subjects with positive hepatitis B core antibody titers and normal liver transaminases are allowed provided that antiviral prophylaxis is administered per institutional guidelines; NOTE: subjects with hepatitis C antibody will be eligible provided that they do not have elevated liver transaminases or other evidence of active hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2025-12-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz S Nowakowski, Principal Investigator — Academic and Community Cancer Research United
Locations (12):
- United States (12):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - State University of New York Upstate Medical University, Syracuse, New York
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (R2-ICE): Patients receive lenalidomide PO daily on days 1-14, rituximab IV on day 1, ifosfamide IV over 24 hours on day 2, carboplatin IV over 1-2 hours on day 2, and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving CMR, PMR, or NMR may receive 2 more cycles per physician discretion. After completion of 2 cycles of R2ICE treatment, patients achieving objective status of CMR, PMR or NMR may proceed to SCT during the event monitoring phase.> > Carboplatin: Given IV>
  > Etoposide: Given IV>
  > Ifosfamide: Given IV>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Lenalidomide: Given PO>
  > Rituximab: Given IV
Period: Overall Study
Arm/Group | Treatment (R2-ICE)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (R2-ICE)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
ECOG PS [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction.
  ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  ECOG = 0 is better. ECOG = 1 is worse.
  Participants
    0 | 17
    1 | 13
Clinical Stage [Count of Participants; unit: Participants] — Stage 1: The cancer affects only one area - either a single organ or a single cluster of lymph nodes.
  Stage 2: The cancer affects two or more areas on the same side of the diaphragm.
  Stage 3: The cancer affects areas on both sides of the diaphragm. Stage 4: The DLBCL has spread to organs outside the lymphatic system, such as the lungs or bones.
  Participants
    1 | 4
    2 | 2
    3 | 6
    4 | 18
Number of Prior Regimens [Count of Participants; unit: Participants]
  1 Prior Regimen | 27
  2 Prior Regimens | 2
  3 Prior Regimens | 1
Histology by Central Pathology Review [Count of Participants; unit: Participants]
  Diffuse large B-cell lymphoma | 30
  Not Diffuse large B-cell lymphoma | 0
CD20 by Central Pathology Review [Count of Participants; unit: Participants]
  Positive | 30
  Negative | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Phase II)
Description: Will be defined as a complete metabolic response or partial metabolic response. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: At 42 days (after 2 courses) of treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Treatment (R2-ICE): Patients receive lenalidomide PO daily on days 1-14, rituximab IV on day 1, ifosfamide IV over 24 hours on day 2, carboplatin IV over 1-2 hours on day 2, and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving CMR, PMR, or NMR may receive 2 more cycles per physician discretion. After completion of 2 cycles of R2ICE treatment, patients achieving objective status of CMR, PMR or NMR may proceed to SCT during the event monitoring phase.
  >
  > Carboplatin: Given IV
  >
  > Etoposide: Given IV
  >
  > Ifosfamide: Given IV
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Lenalidomide: Given PO
  >
  > Rituximab: Given IV
Arm/Group | Treatment (R2-ICE)
Number analyzed (Participants) | 30
proportion of participants | 0.567 [0.374 to 0.745]

2. Secondary Outcome: Proportion of Patients Proceeding to Stem Cell Transplant
Description: Estimated by the number of patients who proceed to transplant divided by
  > the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.
Time Frame: At 42 days of treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (R2-ICE)
Number analyzed (Participants) | 30
proportion of participants | 0.467 [0.283 to 0.657]

3. Secondary Outcome: Complete Metabolic Response Rate
Description: Estimated by the number of patients with an objective status of complete metabolic response divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true complete metabolic response rate will be calculated.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (R2-ICE)
Number analyzed (Participants) | 30
proportion of participants | 0.333 [0.173 to 0.528]

4. Secondary Outcome: Overall Survival
Description: The percentage of participants alive will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (R2-ICE)
Number analyzed (Participants) | 30
percentage of participants | NA [14.4 to NA] — Not enough events of death.

5. Other Pre Specified Outcome: Histologic Subtype (Germinal Center B-cell-like Versus Activated B-cell-like Versus Unclassified Subtype)
Description: Evaluated by 2 methods: Hans algorithm by immunohistochemistry and gene expression profiling using nanostring technology. For each method, the relationship between overall response (responder versus non-responder) complete response rate and subtype will be evaluated using Chi-square tests (or Fisher's exact test if the data in the contingency table is sparse).
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Standardized Uptake Value
Description: Evaluated by calculating the percentage (%) standardized uptake value noted on interim positron emission tomography/computed tomography scan and correlated with the overall response (responder versus non-responder) by using a two sample t-test.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Anatomic Size Reduction
Description: Evaluated by calculating the percentage (%) anatomic size reduction noted on interim positron emission tomography/computed tomography scan and correlated with the overall response (responder versus non-responder) by using a two sample t-test.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Minimum Residual Disease Detection in Blood
Description: The correlation of minimal residual disease detection (positive versus negative) with overall response will be evaluated using Chi-square tests (or Fisher's exact test if the data in the contingency table is sparse).
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Minimum Residual Disease Blood Level
Description: The correlation of minimal residual disease quantification (responder versus non-responder) with overall response will be evaluated using two sample t-tests.
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Serum Sample Collected and Stored for Future and Ongoing Research
Description: Some of the initial work for which this would be utilized would include but not limited to studying the serum free light chains, serum free deoxyribonucleic acid and the minimal residual disease. These measures will be summarized descriptively using medians and ranges (continuous measures) or frequencies (categorical measures).
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Treatment (R2-ICE)
All-Cause Mortality (participants affected / at risk) | 12/30
Serious Adverse Events (participants affected / at risk) | 16/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (R2-ICE) (N=30)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 4 (6)
White blood cell decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (R2-ICE) (N=30)
Anemia (Blood and lymphatic system disorders) | 13 (25)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 8 (9)
Pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 10 (20)
Neutrophil count decreased (Investigations) | 24 (50)
Platelet count decreased (Investigations) | 28 (61)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 24 (57)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (15)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (10)
Flushing (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02628405/Prot_SAP_000.pdf